CLINICAL TRIAL: NCT03166254
Title: Pilot Feasibility Study of the Combination of a Personalized Therapeutic Anti-tumor Vaccine With Pembrolizumab and Standard of Care Chemotherapy in Squamous Non-Small Cell Lung Cancer and Extensive Stage Small Cell Lung Cancer
Brief Title: Personalized Therapeutic Anti-tumor Vaccine With Pembrolizumab and Standard of Care Chemotherapy in Squamous Non-Small Cell Lung Cancer and Extensive Stage Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lost funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-x429
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Non Small Cell Lung Cancer; NSCLC; Non-small Cell Lung Cancer; Small Cell Lung Extensive Stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Biopsy; poly ICLC; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Stage IV squamous NSCLC (Experimental): * 4 cycles of standard of care (SOC) platinum doublet chemotherapy (investigator's choice)
  * Pembrolizumab (200 mg every 3 weeks (Q3W) for 4 cycles while patient is receiving SOC chemo). Pembrolizumab may continue to be administered Q3W for a maximum of 35 total administrations
  * All patients will begin the NEO-PV-01 vaccination at Week 12, 3 weeks following the 4th cycle of pembrolizumab / chemotherapy. At Week 12 (Cycle 5), NEO-PV-01 vaccinations will be administered in a prime-boost schedule with 5 priming vaccinations over a 3 week period followed by booster vaccinations at 1 month and 2 months after the last priming vaccination
  * Up to 20 personalized vaccine peptides will be administered for each patient. Vaccine administration will occur on Days 1, 4, 8, 15 during Cycle 5 of pembrolizumab administration and Day 1 of Cycle 6 of pembrolizumab administration, on Day 8 during Cycle 7 of pembrolizumab administration, and on Day 15 during Cycle 8 of pembrolizumab administration
  Interventions: Drug: Pembrolizumab; Biological: NEO-PV-01 vaccine; Procedure: Biopsy; Drug: Poly ICLC; Procedure: Leukapheresis; Procedure: Peripheral blood samples
- Cohort B: Extensive stage SCLC (Experimental): * 4 cycles of standard of care (SOC) platinum doublet chemotherapy (investigator's choice)
  * Pembrolizumab (200 mg every 3 weeks (Q3W) for 4 cycles while patient is receiving SOC chemo). Pembrolizumab may continue to be administered Q3W for a maximum of 35 total administrations
  * All patients will begin the NEO-PV-01 vaccination at Week 12, 3 weeks following the 4th cycle of pembrolizumab / chemotherapy. At Week 12 (Cycle 5), NEO-PV-01 vaccinations will be administered in a prime-boost schedule with 5 priming vaccinations over a 3 week period followed by booster vaccinations at 1 month and 2 months after the last priming vaccination
  * Up to 20 personalized vaccine peptides will be administered for each patient. Vaccine administration will occur on Days 1, 4, 8, 15 during Cycle 5 of pembrolizumab administration and Day 1 of Cycle 6 of pembrolizumab administration, on Day 8 during Cycle 7 of pembrolizumab administration, and on Day 15 during Cycle 8 of pembrolizumab administration
  Interventions: Drug: Pembrolizumab; Biological: NEO-PV-01 vaccine; Procedure: Biopsy; Drug: Poly ICLC; Procedure: Leukapheresis; Procedure: Peripheral blood samples

INTERVENTIONS:
Drug: Pembrolizumab — -Pembrolizumab will be given intravenously over the course of 30 minutes
  Other Names: Keytruda
Biological: NEO-PV-01 vaccine — -Generation of the vaccine is expected to take approximately 12 weeks
  Other Names: Personalized vaccine
Procedure: Biopsy — -Surgical or core needle biopsy of an accessible site for DNA and RNA sequencing, immunological analysis, and generation of NEO-PV-01 vaccine
Drug: Poly ICLC — -NEO-PV-01 is combined with the adjuvant poly-ICLC prior to administration.
  Other Names: Hiltonol
Procedure: Leukapheresis — -Peripheral blood mononuclear cells (PBMCs) for comprehensive immune system monitoring will be obtained from leukapheresis samples collected up to 7 days prior to initiation of NEO PV-01 vaccination and at 7 days (Week 20) following the first NEO-PV-01 booster vaccination.
Procedure: Peripheral blood samples — -Blood samples (80 mL) for immune monitoring will be obtained prior to study treatment and at Weeks 6, 14, 16, 24, 36, 48, 63, 75, 87, and 99.

SUMMARY:
Both metastatic squamous non-small cell lung cancer (NSCLC) and extensive stage small cell lung cancer (SCLC) are incurable with current therapies, but due to mutations induced by cigarette smoke, typically express a large number of altered proteins that can be recognized as foreign by the immune system. This antigenicity is thought to explain the efficacy of pembrolizumab as either a first or second line treatment in this disease. For patients who receive chemotherapy plus immunotherapy as a first line therapy, there is sound rationale for combination treatment with immunotherapy and a therapeutic antitumor vaccine as a maintenance strategy. Regardless of PD-L1 expression in the tumor, monoclonal antibodies that block PD-1/PD-L1 interactions are effective second line therapies after chemotherapy in both NSCLC and SCLC. In addition, by targeting the immune system against tumor specific antigens using a peptide vaccine, the efficacy of pembrolizumab alone is expected to be enhanced, with an improved response rate and prolonged overall survival with no additional toxicity.

This pilot study will provide a preliminary test of the feasibility of generating a personalized, tumor neoantigen-specific therapeutic vaccine and the safety of combining it with checkpoint blockade immunotherapy.

DETAILED DESCRIPTION:
Please note that this study originally opened with ID# 201707041 but was withdrawn due to change in standard of care chemotherapy. This study was revised and submitted as an amendment to the same IND but our IRB required it to be submitted as a new study and it received a new ID#.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Histologically confirmed stage IV squamous NSCLC
* Cohort B: Histologically confirmed extensive stage SCLC
* Sufficient tumor tissue must be available for histologic assessment of PD-L1 expression and for sequence and immunological analysis.
* Measurable disease by RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* At least 18 years of age on the day of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Normal bone marrow and organ function as defined in the table below within 10 days of study entry:

  * Absolute neutrophil count (ANC): ≥1500/µL
  * Platelets: ≥100 000/µL
  * Hemoglobin: ≥9.0 g/dL or ≥5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks)
  * Creatinine: ≤1.5 × upper limit of normal (ULN) OR
  * Measured or calculated2 creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≥30 mL/min for patient with creatinine levels / >1.5 × institutional ULN
  * Total bilirubin: ≤1.5 ×ULN OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 × ULN
  * AST (SGOT) and ALT (SGPT): ≤2.5 × ULN (≤5 × ULN for patients with liver metastases)
  * International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT): ≤1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Male Patients: A male patient must agree to use a contraception as detailed in this protocol during the treatment period and for at least 120 days, corresponding to time needed to eliminate any study treatment(s) after the last dose of study treatment and refrain from donating sperm during this period.
* Female Patients: A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: A woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatment(s). Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Cohort A: Received any prior systemic therapy for cancer treatment.
* Cohort B: May not have received more than one cycle of platinum doublet given with or without an anti-PD-1 or anti-PD-L1 immunotherapeutic.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to day 1 or who has not recovered (ie, ≤ Grade 1 or at baseline from adverse events due to previous therapies). Patients with ≤Grade 2 neuropathy may be eligible.

Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

* Received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Patients may not receive or have received any radiation therapy at the biopsy sites.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has had an allogeneic tissue/solid organ transplant.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 10 mg prednisone daily or any other form of immunosuppressive therapy within 7 days prior to Day 1.
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Prior treatment with a cancer vaccine.
* Prior treatment with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Received a live vaccine within 30 days prior to Day 1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to Day 1 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.

Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

-Currently receiving any other investigational agents or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to Day 1.

Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, underlying pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids (prednisone dose of 10 mg or less per day is allowed), or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* A woman of childbearing potential who has a positive urine pregnancy test within 72 hours prior to treatment allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority.

* Known history of active tuberculosis (TB).
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of the combined regimen as measured by number of participants who experience a serious adverse event | 30 days following the completion of treatment (estimated to be 2 years and 16 weeks)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.

SECONDARY OUTCOMES:
Objective response rate as measured by RECIST 1.1 | Through completion of treatment (estimated to be 108 weeks)
  --Percentage of participants who experience a complete or partial response
  * Complete Response (CR): Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Progression-free survival (PFS) as measured by RECIST 1.1 | Through completion of follow-up (estimated to be 7 years)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Overall survival (OS) | Through completion of follow-up (estimated to be 7 years)
Clinical benefit rate (CBR) | Through completion of treatment (estimated to be 108 weeks)
Duration of response (DOR) | Through completion of treatment (estimated to be 108 weeks)
Response conversion rate (RCR) | Through completion of treatment (estimated to be 108 weeks)
Objective response rate (ORR) as measured per iRECIST | Through completion of treatment (estimated to be 108 weeks)
Progression-free survival (PFS) as measured per iRECIST | Through completion of follow-up (estimated to be 7 years)
  -PFS is defined as the duration of time from start of personalized vaccine treatment (~12 weeks after baseline) to time of progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu